CLINICAL TRIAL: NCT00707148
Title: Safety and Immunogenicity of Tdap Vaccine in Healthy Pregnant Women, Safety in Their Neonates, and Effect of Maternal Immunization on Infant Immune Responses to DTaP Vaccine
Brief Title: Pertussis Vaccine in Healthy Pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0048; H-19633; HHSN272200800002C
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2012-08

CONDITIONS: Diphtheria; Pertussis; Tetanus
Keywords: pertussis, diptheria, tetanus, vaccine, Tdap
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Group 2: Control (Active Comparator): 16 pregnant women to receive: antepartum: saline; postpartum; Tdap vaccine.
  Interventions: Drug: Placebo; Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed
- Group 1: Intervention (Experimental): 32 pregnant women to receive: antepartum: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed (Tdap) vaccine; postpartum: saline.
  Interventions: Drug: Placebo; Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed
- Group 3: Control (Active Comparator): 32 non-pregnant women to receive a single dose of Tdap vaccine.
  Interventions: Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed

INTERVENTIONS:
Drug: Placebo — Saline (0.9% NaCl) administered as a single 0.5 mL intramuscular injection into the deltoid.
  Arms: Group 1: Intervention; Group 2: Control
Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed — Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine absorbed (Tdap). Administered as a single 0.5 mL intramuscular injection into the deltoid.

SUMMARY:
The purpose of this study is to look at the safety and immunogenicity of a combination vaccine that includes tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis (Tdap). The study will be conducted in 48 pregnant women and 32 non-pregnant women. Safety of the newborn infant and the effect of the mother's vaccination on the infants' immune responses prior to vaccinating infants with another combination vaccine to protect against diphtheria, tetanus, and pertussis will be evaluated. Participants will be 18-45 years old. Pregnant volunteers will be 30-32 weeks pregnant and at a low risk for pregnancy complications. Pregnant volunteers will receive 2 injections (1 vaccine and 1 placebo, inactive substance); non-pregnant volunteers will receive 1 injection of vaccine. Blood samples will be collected from the mother and infant, along with the baby's growth measurements. Participation for mother infant pairs is about 15 months and about 7 months for non-pregnant women.

DETAILED DESCRIPTION:
Pertussis, "whooping cough", caused by the gram negative pleomorphic bacillus, Bordetella pertussis, is a highly contagious, potentially life-threatening respiratory illness that has re-emerged in the United States (US) as a cause of morbidity and mortality in infants less than 6 months of age as well as morbidity in adolescents and adults. Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed (Tdap) immunization of women in the third trimester of pregnancy represents an opportunity to protect the vulnerable very young infants through passively acquired maternal pertussis specific antibodies. Tdap vaccine is being evaluated for this purpose since there is no monovalent acellular pertussis (aP) vaccine available in the U.S. This is a multi-site, randomized, double masked, cross-over study in 48 healthy pregnant women, 18-45 years of age who will be randomized (2:1) into two groups. One group will receive a single dose of Tdap vaccine at 30-32 weeks of gestation and a postpartum dose of saline. The other group will receive saline at 30-32 weeks of gestation and a postpartum dose of Tdap vaccine. On May 30, 2008 the Advisory Committee on Immunization Practices (ACIP) issued a recommendation for use of Tdap in pregnant and postpartum women: "Pregnant women (including women who are breastfeeding) who have not received a dose of Tdap previously should receive Tdap after delivery and before discharge from the hospital or birthing center if 2 years or more have elapsed since the most recent administration of Td." This study design provides a control for the evaluation of the safety of Tdap vaccine administered during pregnancy and provides compliance with the ACIP recommendation. Immune responses to Tdap vaccine measured in antepartum and postpartum women enrolled in this clinical trial will be compared. Also, immune responses of the 32 pregnant women antenatally immunized with Tdap will be compared to those in approximately 32 healthy non-pregnant women contemporaneously enrolled into 2 age groups (18-39 years and 40-45 years) that are equal to the pregnant women. The purpose of this study is to evaluate the safety of Tdap vaccine in pregnant women and their neonates and the effect of maternal immunization on the infant immune response to DTaP vaccinations. The safety of and immune response to Tdap vaccine in the 32 pregnant women immunized antenatally will be compared to that in approximately 32 non-pregnant women enrolled contemporaneously. The primary objectives of this phase I study are: to evaluate the safety of a single 0.5 mL intramuscular injection of Tdap vaccine in healthy pregnant women vaccinated at 30-32 weeks of gestation compared to women immunized postpartum and a non-pregnant control group; and to evaluate the safety of maternal Tdap immunization in neonates. Secondary objectives are: to assess the immunogenicity of Tdap vaccine in healthy pregnant women compared to women immunized postpartum and a non-pregnant control group; to determine the efficiency of placental transport of maternal pertussis specific antibodies to the neonate; to assess the persistence of the maternal pertussis specific antibodies in infants just prior to receiving the first dose of DTaP [Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate] vaccine for infants); and to assess the effects of maternal immunization with Tdap vaccine on infant immune responses to DTaP vaccinations. Study duration will be approximately 3 years. Subject participation will be approximately 15 months (for each mother-infant pair) and 7 months for non-pregnan

ELIGIBILITY:
Inclusion Criteria:

Pregnant subjects must meet all inclusion criteria in order to be eligible to participate in the study.

* 18 - 45 years of age
* In the 30th-32nd week of a pregnancy at low risk for complications as determined by the Obstetrical Risk Assessment Form [ORAF] and the following criteria:

All Pregnant Women:

* Second trimester or later ultrasound with no significant abnormalities.
* Alpha fetal protein (AFP) testing, one of the following:

  1. Normal maternal serum AFP performed at 15-20 weeks' gestation (either as part of the quad screen or separately)
  2. Abnormal maternal serum AFP at 15-20 weeks' gestation followed by an amniocentesis demonstrating no chromosomal abnormalities AND either normal amniotic fluid AFP or normal amniotic fluid acetylcholinesterase (AChE) levels.
  3. If a serum AFP test is not performed, one of the following:

  i. A level II ultrasound with no significant abnormalities ii. A normal amniotic fluid AFP test AND an amniocentesis demonstrating no chromosomal abnormalities must be documented.

Pregnant Women 40-45 years of age: no chromosomal abnormalities identified by diagnostic testing [chorionic villus sampling (CVS) or amniocentesis].

* Pregnant Women 18-39 years of age: at least one of the following:

  1. Level II ultrasound with no significant abnormalities
  2. No chromosomal abnormalities identified by diagnostic testing (CVS or amniocentesis)
  3. Pregnancy estimated to be at low risk (< 1 in 270) for Down's syndrome (trisomy 21), trisomy 13 and trisomy 18 by appropriate first or second trimester screening test. Appropriate screening test includes any one of the following:

  i. first trimester screening (nuchal translucency measurement, pregnancy-associated plasma protein A (PAPP-A), and beta- human chorionic gonadotropin (B-hCG) ii. first trimester screening and second trimester quad screen, with risk estimated using an integrated, sequential, or contingency approach iii. second trimester quad screen alone
* Intend to be available for follow-up visits and phone call access through 13 months following delivery
* Willing to have infant immunized with Pentacel vaccine at 2, 4, 6, and 12 months of age
* Willing to give written informed consent

Non-pregnant subjects must meet all inclusion criteria in order to be eligible to participate in the study.

* 18-39 years of age or 40-45 years of age
* Intend to be available for a follow-up visit and phone call access through 6 months following receipt of Adacel vaccine
* Willing to give written informed consent
* Must fulfill one of the following: (i) she is not able to bear children because she has been surgically sterilized (tubal ligation, bilateral oophorectomy or hysterectomy) for at least one year or is at least 1 year post-menopausal or (ii) she agrees to practice effective methods of contraception including, but not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods, birth control pills, patches or hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices), during the study period between enrollment and 30 days following receipt of the vaccine. (If subject is of childbearing potential, the method of birth control will be documented.)
* For a female subject of childbearing potential, must have a negative pregnancy test (urine or serum) within 24 hours prior to vaccination

Exclusion Criteria:

Pregnant subjects who meet any exclusion criteria at baseline will be excluded from the study.

* Serious underlying medical condition (e.g., immunosuppressive disease or therapy, human immunodeficiency virus (HIV) infection, collagen vascular disease, diabetes mellitus, chronic hypertension, moderate to severe asthma, lung/heart disease, liver/kidney disease, chronic or recurrent infections).
* Significant mental illness (e.g. schizophrenia, psychosis, major depression).
* Currently smoking or using illegal substances.
* History of a febrile illness (greater than or equal to 100.4 degrees Fahrenheit or 38 degrees Celsius) within the past 72 hours for antepartum injection or febrile illness (greater than or equal to 100.4 degrees Fahrenheit or 38 degrees Celsius) within 24 hours for postpartum injection.
* Previous severe reaction to any vaccine.
* Receipt of tetanus-diphtheria toxoid immunization within the past 2 years.
* Receipt of tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine absorbed (Tdap) immunization ever.
* Receipt of a vaccine (excluding influenza), blood product (excluding Rhogam) or experimental medicine within the 4 weeks prior to antepartum injection through 4 weeks following post-partum injection. However, measles-mumps-rubella vaccine is permitted post-partum.
* Receipt of or plans to receive influenza vaccine within the 2 weeks prior to or following antepartum injection.
* Deemed high risk for serious obstetrical complication as determined by the Obstetrical Risk Assessment Form.
* Anything in the opinion of the investigator that would prevent volunteers from completing the study or put the volunteer at risk.

Non-pregnant subjects who meet any exclusion criteria at baseline will be excluded from the study.

* Serious underlying medical condition (e.g., immunosuppressive disease or therapy, HIV infection, collagen vascular disease, diabetes mellitus, chronic hypertension, moderate to severe asthma, lung/heart disease, liver/kidney disease, chronic or recurrent infections).
* Significant mental illness (e.g. schizophrenia, psychosis, major depression).
* Currently smoking or using illegal substances.
* History of a febrile illness (greater than or equal to 100.4 degrees Fahrenheit or 38 degrees Celsius) within the past 24 hours.
* Previous severe reaction to any vaccine.
* Receipt of tetanus-diphtheria toxoid immunization within the past 2 years.
* Receipt of Tdap immunization ever.
* Receipt of or plans to receive an investigational or licensed vaccine (excluding influenza), blood product or experimental medicine within the 4 weeks prior to Adacel vaccination through 4 weeks following Adacel vaccination
* Receipt of or plans to receive influenza vaccine within the 2 weeks prior to or following Adacel vaccination.
* Intends to become pregnant during the study period between enrollment and 30 days following receipt of the vaccine.
* Anything in the opinion of the investigator that would prevent a volunteer from completing the study or put the volunteer at risk.

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of injection site and systemic reactions following injections. | Recorded 0 to 7 days after injection.
Frequency of vaccine-associated adverse events (AEs). | 30 minutes post-injection, Day 0, 1-2, 7, 4 weeks post-injection, delivery, Day 1-2, 7, and 2 and 4 months post-delivery. Infant AEs: Delivery, 2, 4, 7, and 13 months. Non-pregnant: Day 0, 1-2, 7, 4 weeks and 6 months.
Frequency of vaccine-associated serious adverse events (SAEs). | Maternal SAEs through 4 months post delivery and infant SAEs from delivery to 13 months. Non-pregnant SAEs: Day 0 through to 6 months post-injection.
Infant growth measurements (fronto-occipital circumference [FOC], length and weight). | At delivery and at 2, 7 and 13 months of age.
Bayley III developmental screening of infants. | At age 13 months.
Incidence of pertussis infection captured by surveillance for adverse events (AEs) and serious adverse events (SAEs). | Duration of study, captured by surveillance for AEs and SAEs. Antepartum: Day 1-2 and 7; 4 weeks; delivery. Postpartum: Day 1-2 and 7; Month 2, 4,7, and 13.

SECONDARY OUTCOMES:
Concentrations of immunoglobulin G (IgG) for pertussis toxin (PT), pertactin (PRN), fimbrial proteins (FIM), filamentous hemagglutinin (FHA), tetanus toxoid (TT), and diphtheria toxoid (DT). | Mother: blood samples collected before and 4 weeks after antepartum injection, at hospital admission for delivery and at the 2 month post delivery visit. Infant: collected at delivery (cord), 2, 7 and 13 months of age.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Duke University Medical Center - Duke Perinatal Clinic, Durham, North Carolina
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington
  - Seattle Children's Hospital - Infectious Diseases, Seattle, Washington

REFERENCES:
- [Result] Munoz FM, Bond NH, Maccato M, Pinell P, Hammill HA, Swamy GK, Walter EB, Jackson LA, Englund JA, Edwards MS, Healy CM, Petrie CR, Ferreira J, Goll JB, Baker CJ. Safety and immunogenicity of tetanus diphtheria and acellular pertussis (Tdap) immunization during pregnancy in mothers and infants: a randomized clinical trial. JAMA. 2014 May 7;311(17):1760-9. doi: 10.1001/jama.2014.3633. PMID 24794369